CLINICAL TRIAL: NCT03471104
Title: The Use of Patient-Reported Outcome Measures (PROMs) to Promote Quality of Clinical Diabetes Consultations
Brief Title: The Diabetes Patient-Reported Outcome Measures Trial
Acronym: DiaPROM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We have piloted the trial and concluded not to proceed to a fullscale trial.
Sponsor: Haukeland University Hospital (Other)
Collaborators: Western Norway University of Applied Sciences (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2017-01506
Record Dates: First submitted 2018-02-22; First posted 2018-03-20 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes-related distress; Living with diabetes; Patient-Reported Outcome Measures (PROMs)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAID in clinical diabetes consultations (Experimental): Participants randomised to the intervention arm. Participants complete the Problem Area in Diabetes scale (PAID) and evaluation PROMs. Participants with specified PAID scores will be offered an empowerment-based follow-up by diabetes specialist nurses.
  Interventions: Other: PAID in clinical diabetes consultations
- Control group (No Intervention): Participants randomised to the control group. Participants complete PROMs but the results/answers will not be available in the electronic patient records until the trial is finished. The participants will receive standard care.

INTERVENTIONS:
Other: PAID in clinical diabetes consultations — The intervention starts when participants complete PROMs before an annual consultation. The physician reviews the PAID (problem areas in diabetes scale) scores with the participant. Participants with one or more single PAID item(s) scored 3 or 4, or a PAID score ≥30, will be referred to extra follow-up which will consist of at least two diabetes nurse consultations. The nurses will follow a communication manual based on key elements from empowerment theory and self-determination theory.
  The participants then complete the PROMs prior to the next annual consultation with the physician.
  Other Names: DiaPROM
  Arms: PAID in clinical diabetes consultations

SUMMARY:
The study aim to evaluate the use of Patient-Reported Outcome Measures in clinical diabetes consultations.

DETAILED DESCRIPTION:
The psychological and emotional impact of living with diabetes is greatly underreported in clinical diabetes care, and diabetes distress is found to be associated with decreased glycemic control. Therefore, regular assessment of diabetes distress is recommended. The integration of assessments with Patient-Reported Outcome Measures (PROMs) in clinical practice has the potential to enhance care for people with diabetes by identifying problems and improving patient-clinician communication. The overall aim of the DiaPROM trial is to develop, test and evaluate the effectiveness of a structured empowerment-based intervention with the use of a PROM regarding diabetes distress as a tool for needs assessment and dialogue support in clinical diabetes consultations among adults with Type 1 Diabetes. The investigator's hypothesis is that the intervention primarily will reduce diabetes distress and secondarily improve overall well-being, improve the perceived competence for diabetes management, improve glycemic control, and improve satisfaction with the diabetes follow-up.

ELIGIBILITY:
1. Inclusion Criteria:

   * type 1 diabetes for more than one year
2. Exclusion Criteria:

   1. not being able to read and complete questionnaires on the computer because of

      * language problems
      * reading problems
      * cognitive problems
   2. pregnancy
   3. severe somatic and psychiatric co-morbidities

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes Distress Scale (DDS) | Baseline, 12 months and 24 months.
  Self reported diabetes-related distress. 17 items are scored on a 6 point Likert scale from 1 "not a problem" to 6 "very serious problem". Scores are summated and divided by 17 to form a mean/average score. There are also four subscales; emotional burden (5 items), physician-related distress (4 items), regimen-related distress (5 items) and interpersonal distress (3 items). The subscale scores are calculated similar to the total score except for dividing by the number of items for each subscale. A total DDS-score or subscale score of more than 3 is regarded as high degree of diabetes distress. Whilst a score of 2 indicate moderate diabetes distress and a score of 1 is considered as low degree of diabetes distress.

SECONDARY OUTCOMES:
Change in The World Health Organisation 5-wellbeing scale (WHO-5) | Baseline, 12 months and 24 months.
  Self reported emotional wellbeing. 5 items are scored on a 6 point Likert scale from 0 "never" to 5 "all of the time". Scores are summated. Raw score 0 to 25 is transformed to 0-100 by multiplying by 4. Higher values represent better outcome. A score of 50 or below is indicate suboptimal well-being. A score of 28 or below is considered as likely depression.
Change in Perceived Competence for Diabetes Scale (PCDS) | Baseline, 12 months and 24 months.
  Self report of the individuals perceptions of competence for diabetes. 4 items are scored on a 7 point Likert scale from 1 "strongly disagree" to 7 "strongly agree". Scores are summated and divided by 4 to form a mean/average score. Higher score indicate better perceived diabetes competence.
Change in Glycosylated hemoglobin A1c (HbA1c) | Baseline, 12 months and 24 months.
  Blood test: HbA1c refers to glycated hemoglobin, which identifies average plasma glucose concentration. Higher values indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Haugstvedt, PhD, Principal Investigator — Haukeland UH; Marit Graue, PhD, Study Chair — Western Norway University of Applied Sciences; Ragnhild B. Strandberg, PhD, Study Chair — Western Norway University of Applied Sciences; Grethe S. Tell, PhD, Study Chair — University of Bergen; Ingvild Hernar, MSc, Study Chair — University of Bergen, Haukeland UH, Western Norway Uni. of Applied Sciences
Locations (1):
- Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haugstvedt A, Hernar I, Strandberg RB, Richards DA, Nilsen RM, Tell GS, Graue M. Use of patient-reported outcome measures (PROMs) in clinical diabetes consultations: study protocol for the DiaPROM randomised controlled trial pilot study. BMJ Open. 2019 Jan 17;9(1):e024008. doi: 10.1136/bmjopen-2018-024008. PMID 30782722
- [Background] Hernar I, Graue M, Richards DA, Strandberg RB, Nilsen RM, Rekdal M, Lovaas KF, Madsen TV, Tell GS, Haugstvedt A. Use of patient-reported outcome measures (PROMs) in clinical diabetes consultations: the DiaPROM randomised controlled pilot trial. BMJ Open. 2021 Apr 14;11(4):e042353. doi: 10.1136/bmjopen-2020-042353. PMID 33853796
- [Background] Hernar I, Graue M, Strandberg RB, Lie SS, Sigurdardottir AK, Richards DA, Kolltveit BH, Haugstvedt A. Young adults with type 1 diabetes and their experiences with diabetes follow-up and participation in the DiaPROM pilot trial: A qualitative study. Diabet Med. 2021 Jun;38(6):e14535. doi: 10.1111/dme.14535. Epub 2021 Feb 16. PMID 33547702

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03471104/SAP_001.pdf